CLINICAL TRIAL: NCT05834101
Title: Comparative Effects of Myofascial Release and Dynamic Stretching on Flexibility Agility, Jump and Sprint in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0417
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Athletic Injuries
Keywords: Dynamic Stretching Self-Myofascial Release
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofacial Release (Experimental): Illiopsoas , quadriceps, hamstrings, hip adductors, hip abductors ,tensor fasciae lata and gluteus, Foot flexors and extensors received thirty seconds flexibility by foam rolling.Although there appears to be a correlatiomuscle goups between higher SMR length and bigger impact size, the exact link between SMR duration and effect size is uncertain. The time was 30 seconds each muscle group was chosen since it is more realistic than the 60 seconds utilized by MacDonald et al., and it was also used by Peacock et al. Similar to the Grid roller, a commercially available foam roller had net diameter of 12.7 cm and a 5-mm thick empty core of plastic coated with a 12-mm layer of dense foam. In this study, participants were instructed to do the motions in sequenced and save manner, covering the complete muscular area, applying consistent pressure that was felt comfortable. For a total of 16 minutes, the therapy lasted 8 minutes on one leg and 16 minutes on both legs
  Interventions: Other: Myofacial Release
- Dynamic Stretching (Experimental): The regimen included ten dynamic workouts lasting 10 minutes and varying in intensity from medium to high. At a distance of 13 meters, each Dynamic stretching exercise was completed. Before each workout, the subjects were given a 10-second rest time. During the exercises, the participants were given verbal comments on their posture, and video recordings of the activities were displayed to them. Dynamic stretching included High knee walk, Straight-leg march, Hand walk, Lunge walks, Backward lunge, High-knee skip, Lateral shuffle, Back pedal, Heel-ups, and High-knee run
  Interventions: Other: Dynamic streching

INTERVENTIONS:
Other: Myofacial Release — Illiopsoas , quadriceps, hamstrings, hip adductors, hip abductors ,tensor fasciae lata and gluteus, Foot flexors and extensors received thirty seconds flexibility by foam rolling.Although there appears to be a correlatiomuscle goups between higher SMR length and bigger impact size, the exact link between SMR duration and effect size is uncertain. The time was 30 seconds each muscle group was chosen since it is more realistic than the 60 seconds utilized by MacDonald et al., and it was also used by Peacock et al. Similar to the Grid roller, a commercially available foam roller had net diameter of 12.7 cm and a 5-mm thick empty core of plastic coated with a 12-mm layer of dense foam. In this study, participants were instructed to do the motions in sequenced and save manner, covering the complete muscular area, applying consistent pressure that was felt comfortable. For a total of 16 minutes, the therapy lasted 8 minutes on one leg and 16 minutes on both legs
  Arms: Myofacial Release
Other: Dynamic streching — The regimen included ten dynamic workouts lasting 10 minutes and varying in intensity from medium to high. At a distance of 13 meters, each Dynamic stretching exercise was completed. Before each workout, the subjects were given a 10-second rest time. During the exercises, the participants were given verbal comments on their posture, and video recordings of the activities were displayed to them. Dynamic stretching included High knee walk, Straight-leg march, Hand walk, Lunge walks, Backward lunge, High-knee skip, Lateral shuffle, Back pedal, Heel-ups, and High-knee run
  Arms: Dynamic Stretching

SUMMARY:
The study will be a randomized clinical trial. Data was collected from the Pakistan sports board. All 44 Participants were randomly allotted into 2 groups via lottery method, with 22 participants in each group. 10 participants from cricket and volleyball each, 8 from wrestling, athletes, and football each. Participant informed consent was taken priory, and all information was given to them regarding their enrolment in the study. And taken them in confidence that their data was kept confidential and this study does not harm their health. Group A participants received the Myofascial release technique while group B received the dynamic stretching technique. Data were collected pre and post. The session was last for 3 weeks, and each week had 5 sessions. Statistical package for the social sciences will be used to analyze the results by using parametric test after confirming normality of data.

DETAILED DESCRIPTION:
Myofascial treatment aims to stretch and relax the fascia, allowing musculoskeletal structures to move with relaxation and restore the affected individual functionality. This treatment is frequently known as myofascial release therapy. Other people may refer to it as 'myofascial trigger point treatment.

A dynamic warm-up, also known as dynamic stretching, involves using a muscle's force generation and the momentum of the body to increase the range of motion of a joint. A dynamic warm-up is frequently included in a specialized warm-up to make the body get ready for the loads that will be put throughout the game.

Myofascial Release and Dynamic Stretching are different techniques that can be used to Flexibility Agility, Jump and Sprint in the early phase which also lead to an increase in athlete's stability, coordination and build confidence in their performances and limit the incidence of injury.

The physical ability to move musculoskeletal through their full range of motion is known as flexibility. Stretching assists function, and posture, avoid poor body sequence, maintains muscle length, balance, and minimizes the risk of injury The sprint of 40-yard is utilized to evaluate speed, acceleration, and agility. The Agility T-Test is a famous test for assessing athletes' capacity to run forward, reverse, and lateral.

The Vertical leap assessment is used to test an athlete's lower limb strength. sit and reach test used for flexibility of athletes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-35 years.
* No pain complaint
* Recreational activity

Exclusion Criteria:

* joint, meniscus, or ligament damage
* lower extremity surgical history

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Agility T-Test | 3 Months
  To evaluate the athlete's ability to go forward, reverse, and lateral to lateral is mostly by the recognize agility T-test.
Flexibility Sit and Reach Test | 3 Months
  The sit-and-reach method also evaluates the lower limbs with flexibility.The patient reached forward along the measurement line, palms faced downwards and hands were on top of each other or side by side.
Vertical Jump Test | 3 Months
  The Vertical Jump test was used to evaluate an athlete's lower limb strength. A vertical jump test gauge was used.
Sprint Test | 3 Months
  The sprint of 40-yard was used to evaluate an athlete's speed, acceleration, and agility.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- Rashid Usman, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No